CLINICAL TRIAL: NCT07269574
Title: A Multicenter, Retrospective Clinical Study Evaluating the Effect of Different Dietary Patterns on the Prognosis of Ovarian Cancer Patients During PARPi Maintenance Therapy
Brief Title: Impact of Dietary Patterns on Prognosis of Ovarian Cancer Patients During PARPi Maintenance
Status: Not yet recruiting | Type: Observational
Sponsor: Tongji Hospital (Other)
Collaborators: West China Second University Hospital (Other); Peking University People's Hospital (Other); Cancer Hospital Chinese Academy of Medical Science, Shenzhen Center (Other); Union Hospital, Tongji Medical College, Huazhong University of Science and Technology (Other); The Affiliated Hospital of Qingdao University (Other); Qilu Hospital of Shandong University (Other); Shanghai First Maternity and Infant Hospital (Other); First Affiliated Hospital, Sun Yat-Sen University (Other); The First Affiliated Hospital of Soochow University (Other); Henan Provincial People's Hospital (Other); The First Affiliated Hospital of Henan University of Science and Technology (Other); Women's Hospital of Zhejiang University (Unknown); Sun Yat-sen University Cancer Centre (Unknown)
Responsible Party: Principal Investigator, Qinglei Gao, Professor, Tongji Hospital
Other Study IDs: TJH-OVC-PARPi-DIET
Record Dates: First submitted 2025-11-26; First posted 2025-12-08 (Actual); Last update posted 2025-12-08 (Actual); Status verified 2025-11

CONDITIONS: Ovarian Cancer; Fallopian Tube Cancers; Primary Peritoneal Carcinoma; High-grade Serous Ovarian Cancer
Keywords: Ovarian Cancer; High-Grade Serous Ovarian Cancer; PARP Inhibitor; Maintenance Therapy; Dietary Pattern; Low-Carbohydrate Diet
MeSH Terms: conditions — Ovarian Neoplasms; Fallopian Tube Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Biospecimen Retention: Samples With DNA — Venous blood samples (approximately 5 mL) will be collected from consenting participants at the main study center (Tongji Hospital). Samples will be processed into serum/plasma and stored at -80°C for at least 5 years. These biospecimens will be used for analyzing nutritional and metabolic indicators (e.g., albumin, lipids) and conducting exploratory omics research (including metabolomics, proteomics, and/or transcriptomics) to investigate the association between metabolic profiles and PARPi maintenance therapy outcomes.
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Low-Carbohydrate Diet Pattern: Patients with high-grade serous ovarian cancer receiving first-line PARP inhibitor maintenance therapy whose usual dietary carbohydrate intake accounts for a lower proportion of total energy. The primary definition of this group will be patients with a percentage of total energy from carbohydrates below the cohort-specific median, as estimated from the retrospective food frequency questionnaire (FFQ). Alternative cut-offs based on published literature and dietary guidelines will be explored in sensitivity analyses.
- Regular/High-Carbohydrate Diet Pattern: Patients with high-grade serous ovarian cancer receiving first-line PARP inhibitor maintenance therapy whose usual dietary carbohydrate intake accounts for a regular or higher proportion of total energy. The primary definition of this group will be patients with a percentage of total energy from carbohydrates at or above the cohort-specific median, as estimated from the retrospective food frequency questionnaire (FFQ). Alternative cut-offs based on published literature and dietary guidelines will be explored in sensitivity analyses.

SUMMARY:
The goal of this retrospective observational study is to evaluate the relationship between different dietary patterns (specifically low-carbohydrate diets) and the prognosis of patients with high-grade serous ovarian cancer (HGSOC) receiving first-line PARP inhibitor (PARPi) maintenance therapy. The main questions it aims to answer are:

* Is there an association between dietary patterns and patients' Progression-Free Survival (PFS)?
* Is there an association between dietary patterns and Overall Survival (OS)? This is a multicenter, retrospective cohort study. Researchers will review electronic medical records from 14 tertiary hospitals in China to identify women who received first-line PARP inhibitor maintenance for advanced high-grade serous ovarian cancer between 2020 and 2025, and collect information on baseline characteristics, treatments and follow-up outcomes.

Researchers will compare patients with a "low-carbohydrate diet pattern" to those with a "regular/high-carbohydrate diet pattern" to see if there are differences in treatment outcomes and survival.

Participants will:

* Have their clinical, pathological, and treatment data collected from electronic medical records.
* Complete a retrospective Food Frequency Questionnaire (FFQ) via phone or clinic visit to recall their dietary habits during the maintenance treatment period.
* Optionally provide a blood sample for nutrition and metabolic analysis. (For participants at the main study center only) No experimental drugs or specific diets will be given in this study. All anti-cancer treatments are decided by the treating physicians as part of routine clinical care.

ELIGIBILITY:
Inclusion Criteria:

* Female patients aged 18 to <75 years.
* Histologically or cytologically diagnosed with primary high-grade serous ovarian cancer (HGSOC), fallopian tube cancer, or primary peritoneal cancer.
* Received initial tumor cytoreductive surgery (Primary Debulking Surgery or Interval Debulking Surgery) and first-line platinum-based chemotherapy, achieving Complete Response (CR) or Partial Response (PR).
* Received PARP inhibitors as maintenance therapy for the first time following the completion of first-line treatment.
* Complete clinical data available in the electronic medical records, including baseline characteristics, first-line treatment details, PARPi maintenance therapy information, and prognostic follow-up data.
* The patient (or primary caregiver) has normal communication abilities, voluntarily agrees to participate, and is able to cooperate in completing the retrospective Food Frequency Questionnaire (FFQ).

Exclusion Criteria:

* Clinical diagnosis only, without pathological or cytological confirmation.
* Non-high-grade serous histological subtypes (e.g., ovarian clear cell carcinoma, endometrioid carcinoma, mucinous carcinoma, low-grade serous carcinoma).
* Secondary or metastatic ovarian cancer (malignancy originating from other organs).
* Severe deficiency of key clinical or prognostic information that prevents assessment of the primary endpoint.
* Inability to accurately recall dietary information due to cognitive impairment, mental illness, or other reasons.
* Presence of severe metabolic or digestive system diseases during PARPi maintenance therapy that required specific restricted diets (e.g., insulin-dependent diabetes, dialysis-dependent renal insufficiency, short bowel syndrome, active Crohn's disease).
* Occurrence of significant physiological events during the study period that significantly altered dietary structure (e.g., major gastrointestinal surgery).

Ages: 18 Years to 75 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — This study includes only women with ovarian, fallopian tube, or primary peritoneal cancer. These cancers arise in female reproductive organs, so only female patients who have been diagnosed with these conditions and received PARP inhibitor maintenance therapy are eligible for this study.
Study Population: The study population consists of women with primary high-grade serous ovarian cancer, fallopian tube cancer, or primary peritoneal cancer who were treated at 14 tertiary hospitals in China. Eligible patients underwent primary or interval debulking surgery followed by first-line platinum-based chemotherapy, achieved complete or partial response, and then received a PARP inhibitor as first-line maintenance therapy between 2020 and 2025. Participants are identified from hospital electronic medical records, and those who can be contacted and are willing to participate will complete a retrospective food frequency questionnaire about their usual diet during PARP inhibitor maintenance.
Sampling Method: Non-Probability Sample
Enrollment: 600 (Estimated)
Dates: Start 2025-11-27 (Estimated); Primary Completion 2026-11-30 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Progression-Free Survival (PFS) | From the initiation of PARPi maintenance therapy until disease progression or death, assessed up to approximately 60 months (5 years).
  PFS is defined as the duration from the start date of PARP inhibitor (PARPi) maintenance therapy to the date of the first documented disease progression or death from any cause, whichever occurs first. Disease progression is assessed according to Response Evaluation Criteria in Solid Tumors (RECIST) version 1.1 for radiologic progression or Gynecologic Cancer InterGroup (GCIG) criteria for CA-125 biochemical progression.

SECONDARY OUTCOMES:
Overall Survival (OS) | From the initiation of PARPi maintenance therapy until death, assessed up to approximately 60 months.
  OS is defined as the time duration from the start date of PARPi maintenance therapy to the date of death from any cause. For participants who are still alive at the time of data analysis, survival time will be censored at the date of last contact/follow-up.
Duration of PARP Inhibitor Maintenance Therapy | From initiation of PARP inhibitor maintenance therapy to permanent discontinuation or last recorded dose, up to 5 years.
  Duration of PARP inhibitor (PARPi) maintenance therapy is defined as the time from the date of initiation of PARPi maintenance to the date of permanent discontinuation of PARPi for any reason (including disease progression, adverse events, patient preference, financial reasons, or other clinical decisions).
  Participants who are still receiving PARPi at the time of analysis will be censored at the date of the last recorded dose.
  This measure reflects treatment adherence to PARPi maintenance in routine clinical practice.
Rate of Treatment Discontinuation Due to Adverse Events | From the initiation of PARPi maintenance therapy to treatment discontinuation, assessed up to approximately 60 months.
  The percentage of participants who permanently discontinue PARP inhibitor maintenance therapy specifically due to drug-related adverse events or toxicity.

IPD SHARING:
Plan to Share IPD: Undecided
It is currently undecided whether individual participant data (IPD) will be shared. The decision will be subject to compliance with the Data Security Law of the People's Republic of China and regulations on human genetic resources management. At this stage, the study protocol specifies that research results will be reported in aggregated summary forms to protect patient privacy. A final data sharing plan will be determined upon study completion in accordance with applicable laws and institutional policies.